CLINICAL TRIAL: NCT07350902
Title: Impact of Primary Dysmenorrhea on Academic Performance and Quality of Life Among Medical Students at Sohag University
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Fayez Shenouda, Assistant lecturer at Public Health and Community department at Sohag University, Sohag University
Other Study IDs: Soh-Med--25-12-1MD
Record Dates: First submitted 2025-12-21; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Academic performance
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self administered questionnaire — Data will be collected through Self-Administered will be distributed to the students after informed consent from participants, The questionnaire is divided into five sections: -
  1. The first section:
     Information on socio demographic and lifestyle, The survey consisted of inquiries as (sex, age, , marital status, residence, physical exercise, drinking cofee ….)
  2. The second section:
     Including Information on menstrual history:
     - Age at menarche, the regularity of menses, the presence of dysmenorrhea or not……etc.
  3. The third section:
  The WaLIDD questionnaire, namely (Working ability, Location, Intensity, Days of pain)
  The forth section:
  The validated dysmenorrhea and AP impact questionnaire in English was used for the survey The last section is named "DysmenQoL questionnaire" (dysmenorrhea and quality of life) . and it is represented by 20 statements about the negative effects of dysmenorrhea on quality of life

SUMMARY:
Pain is an unpleasant sensation that negatively affects individual experiencing it, depending on its quality, intensity, location, and duration. One of the causes of pain among females is dysmenorrhea. Dysmenorrhea is defined as pain during menstruation. A significant population of females experience mild, moderate or severe pain during menstruation. Primary dysmenorrhea is defined as dysmenorrhea with the absence of any organic pathology starting 6-12 months after the menarche and frequently continuing till menopause, while secondary dysmenorrhea results from gynecologic problems such as adenomyosis, endometriosis, uterine fibroid and others.

DETAILED DESCRIPTION:
In the world, the estimated prevalence of dysmenorrhea ranges from 45% to 93% of women of reproductive age, with adolescents having the highest rates of dysmenorrhea.

Studies suggest that approximately 140 million hours are lost annually from school or work owing to dysmenorrhea. It is a leading cause of recurrent short-term school absenteeism, lack of concentration, no active participation, inability to do homework, failure in an exam, and limitation of activity.

An estimated 15% of adolescent females describe their pain as severe, impacting their quality of life. These adolescents can miss 1 to 3 days of school per menstrual cycle.

Studies have noted that dysmenorrhea can lead to lower academic performance (AP) and poor quality of sleep, resulting in mood changes, such as anxiety and depression

ELIGIBILITY:
Inclusion Criteria:

* • Undergraduate females from the 3 selected faculties in Sohag University

Exclusion Criteria:

* • Students who will refuse to participate in this study.

  * Pregnant females \ females with amenorrhea.
  * Females with gynecological problems as adenomyosis, uterine fibroids and others to exclude secondary dysmenorrhea

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: A cross-sectional survey will be conducted in three randomly chosen faculties' in Sohag University,
  The sample will be selected as follow:
  * 3 medical faculties were selected randomly. [Faculty of Medicine, and faculty of Nursing] medical female students are the study population
  * Students will be selected by stratified random sampling technique.
  * Students from each grade except the first grade will be selected by using random sampling technique after fulfilling the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The WaLIDD questionnaire | December 2027
  The WaLIDD questionnaire contains 4 questions :
  Working ability = 0: never, 1: sometimes, 2: regularly, 3: always; Location = 0: none, 1: 1 location. 2: 2-3 locations, 3: 4 locations; Intensity = 0: never, 1: sometimes, 2: regularly, 3: always; Day of Pain = 0: none, 1: 1-2 days, 2: 3-4 days, 3: more than 5 days So, Each of the four questions is scored from 0 to 3 Total score: The total score ranges from 0 to 12
  The interpretation of the WaLIDD questionnaire is as follows:
  0 = No Dysmenorrhea 1-4 = Mild Dysmenorrhea 5-7 = Moderate Dysmenorrhea 8-12 = Severe Dysmenorrhea
"DysmenQoL questionnaire" (dysmenorrhea and quality of life) | December 2027
  it is represented by 20 statements about the negative effects of dysmenorrhea on quality of life (effects on health and feelings, relationships with family members or friends, couple relationships and professional activity). It consists of twenty statements ,the participants give a score from 1 to 5 for each statement:
  1-"Never"; 2-"Few cases"; 3-"Sometimes"; 4-"Most of the time" ; 5-"Every time".
  We calculate the sum of the scores for each statement and we call it "DysmenQoL score" whose value could vary between 20 and 100. So, high scores indicate low quality of life. The DysmenQoL questionnaire proved to be a reliable and valid method for evaluating the impact of dysmenorrhea on the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Fayez Shenouda, Ass lecturer, Principal Investigator — Faculty of Medicine, Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No